CLINICAL TRIAL: NCT00146601
Title: A Phase II Study of Fulvestrant in Premenopausal Women With Hormone Receptor-Positive Breast Cancer
Brief Title: Fulvestrant in Premenopausal Women With Hormone Receptor-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Lowell General Hospital (Other); Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-075
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Breast Cancer
Keywords: Fulvestrant; Advanced breast cancer; Invasive breast cancer; Stage IV Breast Cancer; Hormone Receptor-Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant

SUMMARY:
The purpose of this study is to test the effectiveness and safety of fulvestrant in premenopausal women with advanced breast cancer.

DETAILED DESCRIPTION:
Patients will receive an injection of fulvestrant on first day of treatment and then again 2 weeks later and again 2 weeks after that. Then patients will receive injections every 4 weeks.

Routine blood tests will be performed each time an injection is given.

Patients will be required to complete a hot flash diary, recording the number and severity of hot flashes they experience on a daily basis.

After every 12 weeks of treatment, patients' disease will be assessed by x-rays or scans. If there is no disease progression, the patient will continue to receive injections every 4 weeks with reassessment every 8 weeks.

Patients will continue to receive treatment as long as there is no disease progression or serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, with stage IV disease.
* Tumors must be positive for estrogen receptors, progesterone receptors, or both.
* Patients must be premenopausal.
* Prior anti-estrogen therapy (with or without ovarian suppression)
* Platelet count > 100,000/mm3
* Age older than 18 years
* ECOG performance status 0-2

Exclusion Criteria:

* Hormonal treatment for metastatic disease
* Pregnant or breast-feeding women
* Postmenopausal
* Concurrent hormonal therapy or chemotherapy
* Prior fulvestrant therapy
* More than three prior chemotherapy regimens for metastatic disease
* Concurrent, long-term anticoagulation therapy
* Severe, uncontrolled intercurrent illness
* History of hypersensitivity to castor oil

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To examine the clinical benefit and response rate of hormone receptor-positive metastatic breast cancer previously treated with anti-estrogen therapy in premenopausal women to treatment with fulvestrant

SECONDARY OUTCOMES:
To determine the safety, time-to-progression, and duration of response for this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Bunnell, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts